CLINICAL TRIAL: NCT04154787
Title: A Randomized, Open-label, Two Arm, Parallel Group, Proof-of-concept Clinical Trial to Investigate the Efficacy and Safety of LNP023 Compared With Rituximab in the Treatment of Subjects With Idiopathic Membranous Nephropathy
Brief Title: Efficacy and Safety of LNP023 Compared With Rituximab in Subjects With Idiopathic Membranous Nephropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023D12201; 2019-001734-34 (EudraCT Number)
Record Dates: First submitted 2019-10-08; First posted 2019-11-06 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Idiopathic membranous nephropathy; MN
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rituximab

STUDY DESIGN:
Masking Description: Open label study for treatment (LNP023 or rituximab).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LNP023 (Experimental): As per protocol V00, participants took LNP023 10 mg orally b.i.d. for 4 weeks followed by LNP023 50 mg orally b.i.d. for 20 weeks.
  As per protocol amendment V01, participants took LNP023 50mg orally b.i.d. for 4 weeks followed by LNP023 200mg for 20 weeks.
  Interventions: Drug: LNP023
- Rituximab (Active Comparator): Rituximab 1 g i.v. at Day 1 and Day 15
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: LNP023 — Investigation of LNP023
  Arms: LNP023
Drug: Rituximab — Comparison of rituximab dose
  Arms: Rituximab

SUMMARY:
This was a randomized, open-label, two arm, parallel group, proof-of-concept, nonconfirmatory study evaluating the efficacy and safety of LNP023 compared with rituximab in subjects with Idiopathic (primary) membranous nephropathy (iMN) who are at high risk of disease progression defined on the basis of anti- Phospholipase A2 Receptor (PLA2R) antibody titer ≥ 60 RU/mL and proteinuria with urine protein (UP) ≥ 3.5 g/24h.

DETAILED DESCRIPTION:
The overall study was planned for a total of 65 weeks and included:

* A screening phase of up to 12 weeks
* A treatment phase of up to 24 weeks
* A post-treatment follow-up period of 29 weeks

As per protocol amendment V01, subjects were randomized 1:1 to LNP023 (investigational drug) or Rituximab (comparator) and followed the below dosing schedule:

* LNP023 50mg orally b.i.d. for 4 weeks followed by 200mg orally b.i.d. for 20 weeks
* Rituximab 1g i.v. infusions on Day 1 and Day 15

Initially, per protocol V00, subjects were planned to be randomized in a 1:1:1 ratio to 3 treatment arms:

* Low dose LNP023: LNP023 10mg orally b.i.d. for 4 weeks followed by 50mg orally b.i.d. for 20 weeks
* High dose LNP023: 25mg orally b.i.d. for 4 weeks followed by 200mg orally b.i.d. for 20 weeks
* Rituximab 1g i.v. infusions on Day 1 and Day 15

Following protocol amendment 1 implementation, ongoing subjects were switched to 200mg b.i.d. dose after their initial 4 weeks of treatment.

3 subjects completed treatment under protocol V00. PK/PD data from the 3 completing subjects under protocol V00 are not included in the study results.

The main reason for protocol amendment V01 was to align with the clinical study results obtained from the interim analysis of ongoing phase 2 trials with LNP023 which had shown a dose dependent inhibition of the complement alternative pathway and support best efficacy results with LNP023 at a dose level of 200mg.

The study was early terminated as LNP023 after interim analysis of 12 LNP023 and 14 rituximab subjects because it could already be predicted at that point that the primary goal of superiority of LNP023 vs rituximab in the reduction of UPCR at 24 weeks was not possible to achieve if the study continued to completion.

ELIGIBILITY:
Inclusion Criteria:

* Female or male adult (≥18 years) subjects at screening visit with a diagnosis of idiopathic (primary) MN confirmed by renal biopsy within 36 months prior to screening. A renal biopsy may be taken at any time during the run-in period to confirm the diagnosis of MN and facilitate subject eligibility, if the most recent biopsy was performed greater than 36 months prior to the screening visit.
* Anti-PLA2R antibody titer of ≥ 60 RU/mL at screening visit. If sites opt to use a local laboratory, with prior agreement with sponsor, an anti-PLA2R titer performed within 4 weeks prior to screening visit can be used.
* Urine protein ≥ 3.5 g/24h at screening and baseline visits
* ≤50% reduction in both anti-PLA2R level and 24h urine protein between screening and baseline
* Estimated GFR (using the CKD-EPI formula) ≥ 30 mL/min per 1.73 m2 at screening
* Receiving stable dose at the maximum recommended dose according to local guidelines or maximum tolerated dose of ACEi and/or ARB and/or statins and/or diuretics for at least 8 weeks prior to Day 1
* Vaccination against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae (in accordance with local guidelines) at least 28 days prior to Day 1 and no longer than 5 years prior to Day 1.

Exclusion Criteria:

* Secondary causes of MN, e.g. systemic autoimmune diseases, solid or haematological malignancies, infections or chronic intake of drugs (e.g. gold salts, NSAIDs, penicillamines)
* Diagnostic renal biopsy showing evidence of crescent formation in glomeruli, suggestive of an alternative or additional diagnosis to primary idiopathic MN.
* Previous treatment with B-cell depleting or B-cell modifying agents such as, but not limited to rituximab, belimumab, daratumomab or bortezomib.
* Previous treatment with immunosuppressive agents such as cyclophosphamide, chlorambucil, mycophenolate mofetil (or equivalent), cyclosporine, tacrolimus or azathioprine within 90 days prior to Day 1. Low dose systemic corticosteroid therapy is permitted, though the subject should have been on stable dose equivalent to ≤10 mg prednisolone for at least 90 days prior to Day 1.
* Previous treatment with gemfibrozil or strong CYP2C8 inhibitors such as clopidogrel within 7 days prior to Day 1
* Presence or suspicion (based on judgment of the investigator) of active infection within 30 days prior to Day 1, or history of severe recurrent bacterial infections
* Known contra-indications for the use of rituximab, including hypersensitivity to the active substance or to murine proteins, or to any of the excipients (sodium citrate, polysorbate 80, sodium chloride, sodium hydroxide, hydrochloric acid, water for injections). Other contra-indications for the use of rituximab, including active, severe infection, patients in a severely immunocompromised state, severe heart failure (NYHA Class IV) or severe, uncontrolled cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-23 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Novartis Investigative Site, Beijing, China
- Novartis Investigative Site, Prague, Czechia
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Jena
- India (2):
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Nijmegen, Netherland, Netherlands
- Spain (2):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Taipei, Taiwan
- United Kingdom (3):
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: CLNP023D12201_NovCTR__28_Dec_2023.docx attachment has been refreshed from the Clinical Trials Results Word Form template. Data may be populated from the following (as available) : Study (123.0), Protocol (9.43), Results(1.6) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217151&parentIdentifier=CLNP023D12201&attachmentIdentifier=69c0c367-eed4-4d39-861b-96ef13c98ed9&fileName=CLNP023D12201_NovCTR__28_Dec_2023.docx&versionIdentifier=
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 18 investigative sites in 9 countries/regions: Argentina (3), Czech Republic (1), Germany (4), India (2), Netherlands (1), Spain (2), United Kingdom (3), China (1) and Taiwan (1)
Groups:
- LNP023 10/50 mg b.i.d.: As per protocol V00, participants took LNP023 10 mg orally b.i.d. for 4 weeks followed by LNP023 50 mg orally b.i.d. for 20 weeks
- LNP023 200 mg b.i.d.: Combination of the LNP023 25/200 mg b.i.d. and 50/200 mg b.i.d. groups. Under protocol V00, participants took LNP023 25 mg orally b.i.d. for 4 weeks followed by LNP023 200 mg orally b.i.d. for 20 weeks.
  Under protocol v01, participants took LNP023 50 mg orally b.i.d. for 4 weeks followed by LNP023 200 mg orally b.i.d. for 20 weeks.
Period: Overall Study
Arm/Group | LNP023 10/50 mg b.i.d. | LNP023 200 mg b.i.d. | Rituximab
Started | 3 | 19 | 15
Completed | 3 | 9 | 14
Not Completed | 0 | 10 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Patient Requires Other Treatment | 0 | 1 | 0
Not completed — Study Terminated By Sponsor | 0 | 6 | 1
Not completed — Subject Decision | 0 | 1 | 0
Not completed — Suspected Lack Of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNP023 10/50 mg b.i.d. | LNP023 200 mg b.i.d. | Rituximab | Total
Number analyzed (Participants) | 3 | 19 | 15 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (18.52) | 48.9 (8.84) | 46.7 (15.33) | 48.5 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 6
  Male | 2 | 15 | 14 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 5 | 4 | 10
  Black Or African American | 0 | 0 | 1 | 1
  Unknown | 0 | 0 | 1 | 1
  White | 2 | 14 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Ratio Between Baseline Urine Protein Creatinine Ratio (UPCR) and Urine Protein Creatinine Ratio at 24 Weeks of Treatment (From 24h Urine Collection)
Description: The primary endpoint of this study is the ratio between UPCR at 24 weeks of treatment measured in 24h urine and baseline UPCR .
  To assess the primary objective, the log-transformed ratio to baseline in UPCR was analyzed using a mixed model for repeated measures (MMRM). The results were back transformed and presented on the original scale.
Time Frame: Baseline, Day 113, Day 169
Population: PD set: In line with the protocol, PD (pharmacodynamics) analyses were performed for all participants who received LNP023 200 mg or rituximab and experienced no protocol deviations with relevant impact on PD/efficacy data. Only participants with a value for UPCR at both Baseline and Day 113 or Day 169 were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio to baseline
Arm/Group | LNP023 200 mg b.i.d. | Rituximab
Number analyzed (Participants) | 10 | 13
ratio to baseline
  Day 113 | 0.94 [0.74 to 1.20] | 0.89 [0.71 to 1.10]
  Day 169: number analyzed (Participants) | 9 | 9
  Day 169 | 0.88 [0.65 to 1.19] | 0.64 [0.48 to 0.86]
Statistical Analysis 1: Comparison: LNP023 200 mg b.i.d. vs Rituximab; Test type: Superiority — Comparison of adjusted geometric mean ratios on Day 169; p = 0.2670, Mixed Models Analysis — Calculated at one-sided 10% level from a lower-tailed test; Adjusted geometric mean ratio = 1.37, 95% CI 2-sided [0.90 to 2.08]

2. Secondary Outcome: Change From Baseline in Plasma Levels of Circulating Fragment of Factor B (Bb)
Description: The drug (LNP023) is expected to block the complement alternative pathway dysregulation and thereby should normalize complement biomarker levels in serum. Bb is a biomarker that accurately reflects the level of complement Alternative Pathway activation.
  Baseline is defined as the last non-missing measurement prior to randomization. Measurements for LNP023 group were done pre-dose.
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 113 and Day 169
Population: PD set: In line with the protocol, PD (pharmacodynamics) analyses were performed for all participants who received LNP023 200 mg or rituximab and experienced no protocol deviations with relevant impact on PD/efficacy data. Only participants with values of plasma levels of circulating fragment of factor B at both Baseline and the different time points were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNP023 200 mg b.i.d. | Rituximab
Number analyzed (Participants) | 17 | 13
ng/mL
  Day 15 | 1520.59 (9370.086) | -417.69 (701.667)
  Day 29: number analyzed (Participants) | 15 | 13
  Day 29 | -732.00 (1412.633) | -318.46 (604.440)
  Day 57: number analyzed (Participants) | 14 | 13
  Day 57 | -545.00 (1379.201) | -75.38 (787.545)
  Day 113: number analyzed (Participants) | 11 | 12
  Day 113 | -877.27 (1562.716) | -219.17 (703.568)
  Day 169: number analyzed (Participants) | 10 | 9
  Day 169 | -984.00 (1794.419) | -570.00 (611.167)

3. Secondary Outcome: Change From Baseline in Plasma Levels of sC5b-9
Description: Soluble C5b-9 (sC5b-9) is a biomarker of the complement pathway activity that correlate with disease progression.
  Baseline is defined as the last non-missing measurement prior to randomization. Measurements for LNP023 group were done pre-dose.
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 113, Day 169
Population: PD set: In line with the protocol, PD (pharmacodynamics) analyses were performed for all participants who received LNP023 200 mg or rituximab and experienced no protocol deviations with relevant impact on PD/efficacy data. Only participants with a value of plasma levels of sC5b-9 at both Baseline and the different time points were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNP023 200 mg b.i.d. | Rituximab
Number analyzed (Participants) | 17 | 13
ng/mL
  Day 15 | -80.40 (98.229) | -38.49 (52.258)
  Day 29: number analyzed (Participants) | 15 | 13
  Day 29 | -82.80 (118.338) | -24.51 (94.826)
  Day 57: number analyzed (Participants) | 14 | 13
  Day 57 | -90.62 (108.483) | -14.02 (107.651)
  Day 113: number analyzed (Participants) | 11 | 12
  Day 113 | -113.32 (108.118) | -24.95 (128.721)
  Day 169: number analyzed (Participants) | 10 | 9
  Day 169 | -84.07 (96.045) | -21.76 (122.654)

4. Secondary Outcome: Ratio to Baseline of Urine Protein Creatinine Ratio (UPCR) Measured in First Morning Void
Description: Adjusted geometric mean ratio to baseline of Urine Protein Creatinine Ratio (UPCR) measured in first morning void.
  First morning void urine sample was collected in the morning of the day before the visit and kept in the fridge.
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 266 and Day 378
Population: PD set: In line with the protocol, PD (pharmacodynamics) analyses were performed for all participants who received LNP023 200 mg or rituximab and experienced no protocol deviations with relevant impact on PD/efficacy data. Only participants with a value of UPCR measured in first morning void at the different time points were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio to baseline
Arm/Group | LNP023 200 mg b.i.d. | Rituximab
Number analyzed (Participants) | 18 | 13
ratio to baseline
  Day 15: number analyzed (Participants) | 15 | 11
  Day 15 | 0.94 [0.65 to 1.34] | 1.15 [0.75 to 1.76]
  Day 29: number analyzed (Participants) | 18 | 12
  Day 29 | 0.98 [0.70 to 1.36] | 0.90 [0.60 to 1.35]
  Day 57: number analyzed (Participants) | 14 | 12
  Day 57 | 1.02 [0.71 to 1.48] | 0.77 [0.51 to 1.16]
  Day 85: number analyzed (Participants) | 11 | 13
  Day 85 | 1.03 [0.68 to 1.56] | 0.75 [0.50 to 1.13]
  Day 113: number analyzed (Participants) | 10 | 11
  Day 113 | 1.05 [0.68 to 1.63] | 0.92 [0.60 to 1.41]
  Day 141: number analyzed (Participants) | 10 | 9
  Day 141 | 0.75 [0.48 to 1.19] | 0.77 [0.48 to 1.23]
  Day 169: number analyzed (Participants) | 9 | 9
  Day 169 | 0.72 [0.44 to 1.16] | 0.55 [0.34 to 0.89]
  Day 266: number analyzed (Participants) | 6 | 7
  Day 266 | 0.57 [0.33 to 0.99] | 0.34 [0.20 to 0.57]
  Day 378 (End Of Study): number analyzed (Participants) | 8 | 8
  Day 378 (End Of Study) | 0.37 [0.22 to 0.63] | 0.46 [0.27 to 0.76]
Statistical Analysis 1: Comparison: LNP023 200 mg b.i.d. vs Rituximab; Day 15; Test type: Superiority; p = 0.4598, Mixed Model for Repeated Measures — Calculated from a two-sided test at the 0.05 significance level; Adjusted geometric mean ratios = 0.81, 95% CI 2-sided [0.47 to 1.42] — Comparison of adjusted geometric mean ratios: Test vs Ref
Statistical Analysis 2: Comparison: LNP023 200 mg b.i.d. vs Rituximab; Day 169; Test type: Superiority; p = 0.4528, Mixed Model for Repeated Measures — Calculated from a two-sided test at the 0.05 significance level; Geometric mean ratios = 1.30, 95% CI 2-sided [0.65 to 2.61] — Comparison of adjusted geometric mean ratios: Test vs Ref

5. Secondary Outcome: Number of Participants by Treatment Response at 24 Weeks of Treatment
Description: Participants were considered complete responders if at 24 weeks of treatment, they showed complete remission of proteinuria (i.e., Urine Protein (UP) ≤ 0.3 g/24h), partial responders if they showed partial remission (i.e., UP > 0.3g/24h and ≤ 3.5 g/24h and a reduction of UP by >50% from baseline), and non-responders if UP >3.5g/24h and/or reduction of UP from baseline <50%.
Time Frame: Baseline, Day 169
Population: PD set: In line with the protocol, PD (pharmacodynamics) analyses were performed for all participants who received LNP023 200 mg or rituximab and experienced no protocol deviations with relevant impact on PD/efficacy data. Only participants with UP values at both baseline and Day 169 were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | LNP023 200 mg b.i.d. | Rituximab
Number analyzed (Participants) | 9 | 9
Participants
  Complete | 0 | 0
  Partial | 2 | 2
  No response | 7 | 7

6. Secondary Outcome: Change From Baseline in (eGFR) Estimated Glomerular Filtration Rate Over Time
Description: Changes in renal function were assessed via estimated glomerular filtration rate (eGFR).
  Change in eGFR was calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: PD set: In line with the protocol, PD (pharmacodynamics) analyses were performed for all participants who received LNP023 200 mg or rituximab and experienced no protocol deviations with relevant impact on PD/efficacy data. Only participants with a eGFR value at both Baseline and the different time points were included in the analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | LNP023 200 mg b.i.d. | Rituximab
Number analyzed (Participants) | 19 | 13
mL/min/1.73 m^2
  Day 15: number analyzed (Participants) | 18 | 13
  Day 15 | 2.3 (12.07) | 0.3 (8.33)
  Day 29 | -0.5 (8.53) | 6.1 (10.44)
  Day 57: number analyzed (Participants) | 14 | 13
  Day 57 | 2.0 (11.10) | 9.2 (21.05)
  Day 85: number analyzed (Participants) | 12 | 13
  Day 85 | -1.6 (11.53) | 10.2 (16.40)
  Day 113: number analyzed (Participants) | 11 | 11
  Day 113 | 1.2 (8.64) | 10.8 (15.41)
  Day 141: number analyzed (Participants) | 10 | 9
  Day 141 | -1.8 (9.10) | 7.1 (9.29)
  Day 169: number analyzed (Participants) | 10 | 9
  Day 169 | -1.3 (7.36) | 3.1 (13.21)

7. Secondary Outcome: Pharmacokinetic Parameter Tmax in Plasma
Description: Pharmacokinetics of LNP023 : Tmax is the time to reach maximum (peak) plasma drug concentration after dose administration (time).
  Actual sampling time points were considered for the calculation of PK parameters.
Time Frame: Day 29 and Day 113 (pre-dose and 0.25 hours, 0.5 hours, 1 hour 2 hours, 4 hours and 6 hours post dose)
Population: PK set: PK (pharmacokinetic) analysis set included all participants with at least one available valid PK concentration measurement, who received any LNP023 and experienced no protocol deviations with relevant impact on PK data. Only participants with PK values at the different time points were included in the analysis.
Measure: Median (Full Range); unit: hours
Groups:
- LNP023 10 mg b.i.d.: Low dose of LNP023 under Protocol V00, LNP023 10mg taken orally b.i.d. during the first 4 weeks of treatment
- LNP023 25 mg b.i.d.: High dose of LNP023 under Protocol V00, LNP023 25mg taken orally b.i.d. during the first 4 weeks of treatment
- LNP023 50 mg b.i.d. (4-week Administration): Under Protocol V01, LNP023 50mg taken orally b.i.d. during the first 4 weeks of treatment
- LNP023 50 mg b.i.d. (20-week Administration): Under Protocol V00, LNP023 50mg taken orally b.i.d. during the last 20 weeks of treatment
- LNP023 200 mg b.i.d.: Under protocol V00, participants took LNP023 25 mg orally b.i.d. for 4 weeks followed by LNP023 200 mg orally b.i.d. for 20 weeks.
  Under protocol v01, participants took LNP023 50 mg orally b.i.d. for 4 weeks followed by LNP023 200 mg orally b.i.d. for 20 weeks.
Arm/Group | LNP023 10 mg b.i.d. | LNP023 25 mg b.i.d. | LNP023 50 mg b.i.d. (4-week Administration) | LNP023 50 mg b.i.d. (20-week Administration) | LNP023 200 mg b.i.d.
Number analyzed (Participants) | 2 | 3 | 10 | 2 | 7
hours
  Day 29: number analyzed (Participants) | 2 | 3 | 10 | 0 | 0
  Day 29 | 2.04 [2.00 to 2.08] | 2.00 [1.00 to 4.00] | 2.03 [1.00 to 4.38] |  |
  Day 113: number analyzed (Participants) | 0 | 0 | 0 | 2 | 7
  Day 113 |  |  |  | 2.05 [2.00 to 2.10] | 1.00 [0.250 to 6.00]

8. Secondary Outcome: Pharmacokinetic Parameter Cmax in Plasma
Description: Pharmacokinetics of LNP023: Cmax is the maximum (peak) observed plasma drug concentration after dose administration (mass x volume-1)
Time Frame: Day 29 and Day 113 (pre-dose and 0.25 hours, 0.5 hours, 1 hour 2 hours, 4 hours and 6 hours post dose)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNP023 10 mg b.i.d. | LNP023 25 mg b.i.d. | LNP023 50 mg b.i.d. (4-week Administration) | LNP023 50 mg b.i.d. (20-week Administration) | LNP023 200 mg b.i.d.
Number analyzed (Participants) | 2 | 3 | 10 | 2 | 7
ng/mL
  Day 29: number analyzed (Participants) | 2 | 3 | 10 | 0 | 0
  Day 29 | 1200 (799) | 2070 (938) | 2140 (917) |  |
  Day 113: number analyzed (Participants) | 0 | 0 | 0 | 2 | 7
  Day 113 |  |  |  | 1220 (304) | 4810 (2850)

9. Secondary Outcome: Pharmacokinetic Parameter AUClast in Plasma
Description: Pharmacokinetics of LNP023: AUClast is the AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1)
Time Frame: Day 29 and Day 113 (pre-dose and 0.25 hours, 0.5 hours, 1 hour 2 hours, 4 hours and 6 hours post dose)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LNP023 10 mg b.i.d. | LNP023 25 mg b.i.d. | LNP023 50 mg b.i.d. (4-week Administration) | LNP023 50 mg b.i.d. (20-week Administration) | LNP023 200 mg b.i.d.
Number analyzed (Participants) | 2 | 3 | 10 | 2 | 7
hr*ng/mL
  Day 29: number analyzed (Participants) | 2 | 3 | 10 | 0 | 0
  Day 29 | 5970 (4150) | 8140 (3080) | 9920 (3960) |  |
  Day 113: number analyzed (Participants) | 0 | 0 | 0 | 2 | 7
  Day 113 |  |  |  | 5940 (989) | 22200 (15600)

10. Secondary Outcome: Pharmacokinetic Parameter AUCtau in Plasma
Description: Pharmacokinetics of LNP023 : AUCtau is the AUC calculated to the end of a dosing interval (tau) at steady-state (amount x time x volume-1)
Time Frame: Day 29 and Day 113 (pre-dose and 0.25 hours, 0.5 hours, 1 hour 2 hours, 4 hours and 6 hours post dose)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LNP023 10 mg b.i.d. | LNP023 25 mg b.i.d. | LNP023 50 mg b.i.d. (4-week Administration) | LNP023 50 mg b.i.d. (20-week Administration) | LNP023 200 mg b.i.d.
Number analyzed (Participants) | 2 | 3 | 10 | 2 | 7
hr*ng/mL
  Day 29: number analyzed (Participants) | 2 | 3 | 10 | 0 | 0
  Day 29 | 9850 (5790) | 12800 (3490) | 16500 (5920) |  |
  Day 113: number analyzed (Participants) | 0 | 0 | 0 | 2 | 7
  Day 113 |  |  |  | 10700 (1640) | 36800 (26100)

11. Secondary Outcome: Pharmacokinetics in Urine: Renal Plasma Clearance Derived From 24 Hour Urine Sample
Description: Pharmacokinetics of LNP023 in urine: Renal plasma clearance derived from 24 hour urine sample
Time Frame: Day 113
Population: PK set: PK (pharmacokinetic) analysis set included all participants with at least one available valid PK concentration measurement, who received any LNP023 and experienced no protocol deviations with relevant impact on PK data. Only participants with PK values at Day 113 were included in the analysis.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | LNP023 50 mg b.i.d. (20-week Administration) | LNP023 200 mg b.i.d.
Number analyzed (Participants) | 1 | 7
L/hr | 0.602 | 1.19 (0.668)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 29 weeks post treatment, up to maximum duration of 53 weeks.
Description: The LNP023 200mg group is the sum of subjects from v00 (25/200mg, n=4) and v01 (50/200mg, n=15). A separation by subgroup was not justified as Part A doses were similar (25 vs 50mg), short-termed (4 weeks) and below levels expected to be efficacious, while the Part B dose of 200 mg was the same for all for up to 20 weeks. Moreover, if separated, the difference in subject numbers may have carried a risk of under- or over-interpretation of findings
Groups:
- Pooled LNP023: Combination of the LNP023 10/50 mg b.i.d., 25/200 mg b.i.d. and 50/200 mg b.i.d. groups.
- Total: Total
Arm/Group | LNP023 10/50 mg b.i.d. | LNP023 200 mg b.i.d. | Pooled LNP023 | Rituximab | Total
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/19 | 0/22 | 0/15 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/19 | 3/22 | 4/15 | 7/37
Other Adverse Events (participants affected / at risk) | 2/3 | 13/19 | 15/22 | 7/15 | 22/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 10/50 mg b.i.d. (N=3) | LNP023 200 mg b.i.d. (N=19) | Pooled LNP023 (N=22) | Rituximab (N=15) | Total (N=37)
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 10/50 mg b.i.d. (N=3) | LNP023 200 mg b.i.d. (N=19) | Pooled LNP023 (N=22) | Rituximab (N=15) | Total (N=37)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 2 | 2 | 0 | 2
Influenza like illness (General disorders) | 0 | 1 | 1 | 0 | 1
Oedema (General disorders) | 0 | 1 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 2 | 2 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 3 | 3 | 1 | 4
Coronavirus infection (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Ear infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Liver function test increased (Investigations) | 0 | 1 | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 3
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 2
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 0 | 2
Headache (Nervous system disorders) | 0 | 3 | 3 | 0 | 3
Hypersomnia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Per protocol, participants randomized to the former LNP023 low dose arm (LNP023 10/50 mg b.i.d.) were included in the safety and PK analyses but not in the PD/efficacy analyses as the low number of subjects would not have allowed for a meaningful analysis and interpretation of PD/efficacy data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT04154787/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT04154787/SAP_001.pdf